CLINICAL TRIAL: NCT03028584
Title: Feasibility of Delivering Electronic Health Record (EHR)-Based Survivorship Care Plans and Planning to Cancer Survivors in a Community Oncology Practice
Brief Title: Survivorship Care Plans in a Community Oncology Practice
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: UW16029; P30CA014520 (NIH); 2016-0760 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2016-11-10; First posted 2017-01-23 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer; Prostate Cancer; Colorectal Cancer
Keywords: BrCa; PrCa; CRCa
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Clinicians: Observe up to N=10 clinicians. Observations will include:
  1. Oncology history and care plan development by clinicians including use of EHR technology to develop care plans and methods used to secure necessary information for care plan creation
  2. Provision and coordination of survivorship care occurring during care team meetings, discussions among clinicians, and survivor visits with clinicians, especially visits in which a care plan is provided to a survivor
  3. Clinician seeking survivorship related information or resources through use of technology or discussion with other clinicians
  4. Survivorship work or tasks performed by the clinician including adding, modifying or extracting information from the EHR and adding or modifying information in the care plan
  Interventions: Behavioral: Survey
- Clinicians and Patients: Surveys of N=30 breast cancer, colon cancer, and prostate cancer patients. Subjects will complete 1st survey electronically in-clinic. Subjects will either be e-mailed or mailed a survey at 4 weeks.
  Survey of clinicians will be sent via e-mail.
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — Subjects (cancer patients and clinicians) will complete up to 2 surveys.

SUMMARY:
This is a two part observational study evaluating the feasibility of implementing an EHR-based model within a community oncology practice.

DETAILED DESCRIPTION:
Part 1: The research team will use a sociotechnical work systems model, developed by researchers at the University of Wisconsin (UW) Systems Engineering Initiative for Patience Safety (SEIPS), to guide analysis of the work system barriers and facilitators to implementing an EHR-based care planning model in community oncology practice, collected from direct observations.

Part 2: The research team will measure reach/maintenance (percentage of survivors with EHR-based survivorship care plans (SCPs) over a 9-month time period) and impact (pre/post survey of patient satisfaction and perceived care coordination).

ELIGIBILITY:
Inclusion Criteria:

* Clinicians: Provide cancer care to BrCa, CRCa or PrCa
* Clinicians: Are a physician, advanced practice practitioner, nurse, or equivalent
* Patients: Have a diagnosis of breast, colorectal, or prostate cancer for which and EHR-based SCP will be provided
* Patients: Have been treated with curative intent (e.g. surgery, chemotherapy and/or radiation therapy) for a Stage 1-3 cancer diagnosis
* Patients: Have received some part of active cancer treatment
* Patients: Have complete active treatment (defined as surgery, chemotherapy, and/or radiation therapy). HER2-based and endocrine therapies may be ongoing and do NOT need to have been completed

Exclusion Criteria:

* Unable to complete or unwilling to answer questions in English
* Patients: Received all active cancer treatment elsewhere (e.g. "observation - only" patients)
* Patients: Have metastatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinicians who provide care for breast, colon, or prostate patients.
  Cancer patients/survivors of breast cancer (BrCa), prostate (PrCa), or colorectal (CRCa) cancer.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
EHR-based SCPs and care planning | Up to 2 years
  Asses whether barriers to EHR-based SCPs and care planning have been mitigated, based on clinician survey.

SECONDARY OUTCOMES:
Feasibility of providing EHR-based care planning, measured by SCP provision rates | Up to 2 years
  Measured by SCP provision rates (percentage of survivors with EHR-based SCPs)
Feasibility of providing EHR-based care planning, measured by the EHR | Up to 2 years
  Measured by survivor access to SCPs, per the EHR
Self-reported change in satisfaction, using survey | Up to 2 years
  The impact of providing EHR-based care planning measured in change of satisfaction with perceived care coordination (assessed prior to and at 4 weeks after SCP provision)
Impact of providing EHR-based care planning | Up to 2 years
  Measured by reported SCP usability, usefulness, and content (assessed prior to and at 4 weeks after SCP provision)

CONTACTS AND LOCATIONS:
Overall Officials: Amyé Tevaarwerk, MD, Principal Investigator — University of Wisconsin, Madison; Mary Sesto, PT, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Cancer Center at ProHealth Care, Waukesha, Wisconsin, United States

REFERENCES:
- See also: UW Carbone Cancer Center Home Page — https://cancer.wisc.edu/